CLINICAL TRIAL: NCT04051021
Title: The Impact of Non-Pharmacological Interventions on Patient Experience, Opioid Use, and Healthcare Utilization in Adult Cardiac Surgery Patients
Brief Title: Non-Pharmacological Interventions on Patient Experience and Healthcare Utilization in Adult Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Julie Piazza, Project Manager, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00161399
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Cardiac Surgery
Keywords: Surgery; Cardiac; Opioids; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Masking Description: Research assistants consenting patients and collecting and analyzing data will be blinded to the allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Other)
  Interventions: Other: Usual Care
- Comfort Coach (Experimental)
  Interventions: Behavioral: Comfort Coach

INTERVENTIONS:
Behavioral: Comfort Coach — A trained comfort coach will provide emotional and psychological interventions at six time points: preoperative clinic, day of surgery, extubation, chest tube removal, discharge, 30-day clinic follow-up, and 90-day post-discharge. Patients will also complete surveys at specific time points (preoperative clinic, hospital discharge, 30-day clinic follow-up, and 90-day post-discharge).
  Arms: Comfort Coach
Other: Usual Care — Patients will complete surveys at specific time points (preoperative clinic, hospital discharge, 30-day clinic follow-up, and 90-day post-discharge).
  Arms: Usual Care

SUMMARY:
This study will assess whether non-pharmacological interventions by a comfort coach affect the amount of opioid pain medication used, as well as perceived physical pain and emotional anxiety and healthcare utilization for adult cardiac surgery patients. Participants that are eligible for the study will be randomized to the comfort coach arm or standard of care. Both groups will complete surveys at the specific time frames in order to compare their outcomes. The study hypothesis is that there will be a decrease in opioid use in the intervention group compared to the standard of care arm during the 90-day perioperative course, as well as a decrease in pain and anxiety along with a lower composite outcome of healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* Receiving a first-time elective status open heart cardiac surgery procedure in the Frankel Cardiovascular Center at Michigan Medicine during the recruitment period through a full or miniature sternotomy incision
* Opioid-naïve, defined as not taking a home opioid medication at time of preoperative H&P

Exclusion Criteria:

* Patients undergoing cardiac transplantation, implantation of ventricular assist device, reoperation, and any planned use of circulatory arrest
* Chronic opioid users defined as taking an opioid at time of preoperative clinic visit
* Non-English speaking
* Inability to understand or complete surveys
* Pregnancy
* Unable to sign legal consent form (legal guardian signature not acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-11-08 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Number of days spent at home within the first 30 days after surgery | up to 30 days after surgery
  Number of days spent at home compared between groups
Number of days in the hospital after surgery | average 5-7 days
Number of days admitted to an extended care facility after discharge from the hospital | up to 30 days after surgery
Number of emergency room visits after discharge from the hospital | up to 30 days after surgery
Number and length of readmissions to the hospital following initial discharge after surgery | up to 30 days after surgery

SECONDARY OUTCOMES:
Brief pain inventory (short) | hospital discharge (within 48 hours of time of hospital discharge)
  This is a 9-question inventory which assesses both pain intensity (sensory dimension) and the interference (reactive dimension) of pain in daily activities. Pain intensity is measured on a 0 - 10 scale, with 0 being no pain and 10 being worst possible.
Postoperative Opioid and Pain Management Questionnaire | approximately 30 days after discharge
  This is an 11-item questionnaire collecting data on opioids prescribed, opioids used, pain scores, opioid storage and disposal practices, and assessment of opioid education.
Picker Patient Experience Questionnaire (PPE-15) | approximately 30 days after discharge
  This is a 15-item questionnaire designed to capture the patient's inpatient experience.
  Each response will be categorized as a problem or non-problem and reported as the percent of respondents reporting a problem, averaged across all PPE-15 domains.
Generalized Anxiety Disorder Scale (GAD-7) | up to approximately 90 days after discharge
  This is a self-administered patient questionnaire with 7 items that measures generalized anxiety disorder. Through a 4-point Likert scale from 'not at all' to 'nearly every day', it is asked how often the patient has been bothered by any of the presented problems. The GAD-7 index is obtained by adding the scores from the questionnaire, after having assigned 0 to the least severe situation, 3 to the most severe one, and 1 and 2 to the intermediate ones. The cut off points 5, 10 and 15 allow to classify the anxiety as none/normal (0-4), mild (5-9), moderate (10-14), and severe (15-21). This will be completed at 4 different times in every patient, ranging from preoperative clinic through 90 (+/-7) day follow up.
Patient Health Questionnaire (PHQ-9) | up to approximately 90 days after discharge
  This is a self-administered instrument that will be used to measure depression in each subject. The PHQ-9 score can range from 0-27 with each of the 9 items can be scored from 0-3 corresponding to "no at all", "several days", "more than half the days" and "nearly every day" responses, respectively. This will be completed at 4 different times in every patient, ranging from preoperative clinic through 90 (+/-7) day follow up
Impact of Events Scale-Revised (IES-R) | approximately 30 days after discharge
  This is a 22-item self-report questionnaire measuring post traumatic stress disorder symptoms. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The IES-R yields a total score ranging from 0 (not at all) to 88 (extremely).
Change in the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | preoperative clinic visit, approximately 30 days after discharge
  This a 12-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The KCCQ-12 clinical summary score is a composite assessment of physical limitations and total symptom scores. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Piazza, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brescia AA, Piazza JR, Jenkins JN, Heering LK, Ivacko AJ, Piazza JC, Dwyer-White MC, Peters SL, Cepero J, Brown BH, Longi FN, Monaghan KP, Bauer FW, Kathawate VG, Jafri SM, Webster MC, Kasperek AM, Garvey NL, Schwenzer C, Wu X, Lagisetty KH, Osborne NH, Waljee JF, Riba M, Likosky DS, Byrnes ME, Deeb GM. The Impact of Nonpharmacological Interventions on Patient Experience, Opioid Use, and Health Care Utilization in Adult Cardiac Surgery Patients: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2021 Feb 16;10(2):e21350. doi: 10.2196/21350. PMID 33591291